CLINICAL TRIAL: NCT00497744
Title: Research Study on the Pharmacokinetic Profile of Intraperitoneal Cefepime in Patients With Continuous Ambulatory Peritoneal Dialysis (CAPD) Peritonitis
Brief Title: A Pharmacokinetic Study of Cefepime After Administration Into Dialysate in Patients With Continuous Ambulatory Peritoneal Dialysis (CAPD) Peritonitis
Status: Completed | Type: Observational
Sponsor: Hospital Authority, Hong Kong (Other Government)
Other Study IDs: KW/EX/05-020; HARECCTR0500027
Record Dates: First submitted 2007-07-06; First posted 2007-07-09 (Estimated); Last update posted 2011-06-16 (Estimated); Status verified 2011-06

CONDITIONS: Peritonitis
Keywords: CAPD peritonitis; Peritoneal Dialysis, Continuous Ambulatory
MeSH Terms: conditions — Peritonitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

INTERVENTIONS:
Drug: Intraperitoneal Cefepime

SUMMARY:
Cefepime is a broad-spectrum antibiotic used in treating CAPD peritonitis. However, medical knowledge has been lacking with regard to its pharmacokinetic profile after it has been administered intraperitoneally. The current study aims at determining the drug level at different time after the drug has been added into the peritoneal fluid in patients with CAPD peritonitis. The results of this study will finally leads to rational prescription of this drug at correct dosages.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years & has been put on CAPD for >= 4 weeks before entering into the study

Exclusion Criteria:

* Known hypersensitivity to cefepime or other cephalosporin; CAPD peritonitis <= 28 days before being enrolled into the study
* Antibiotic treatment within 1 week prior to entry into the study
* Severe exit site or tunnel infection on the day of presentation
* Any conditions that prompt early removal of Tenckhoff catheter irrespective of clinical response to antibiotic treatment
* Abdominal malignancy; Any surgical causes of peritonitis
* Suspected or known fungal or tuberculous peritonitis
* History of dementia or known mental incompetency

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 4 males and 2 females, of age 57.83 +/-11.63 years with urinary creatinine clearance of 0.87+/-2.06ml/min/1.73m2 and admitted for CAPD peritonitis were enrolled. After collection of peritoneal dialysate for cell count and microbiological work-up, all subjects were loaded with 2g cefepime IP and dwelled for 6 hours. This was followed by 250mg cefepime in each subsequent 6-hourly peritoneal dialysis exchange. Plasma cefepime levels were determined at time 0, 1, 2, 4, 8, 12, 16, 24, 48, 72, 96, 120 hrs. Pharmacokinetic analyses were then performed.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Estimated)
Dates: Start 2005-11; Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sze Kit Yuen, Dr, Principal Investigator — Department of Medicine and Geriatrics, Caritas Medical Centre
Locations (2):
- China (2):
  - Caritas Medical Centre, Hong Kong
  - Princess Margaret Hospital, Hong Kong